CLINICAL TRIAL: NCT01917695
Title: Randomised Phase III Clinical Trial on Concurent Chemoradiation vs. Neoadjuvant Chemoradiation and Surgery vs. Neoadjuvant Chemotherapy and Surgery in Early Stage Bulky Cervical Cancers (FIGO Stages IB2, IIA2 and IIB)
Brief Title: Study on Early Stage Bulky Cervical Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajkumar Kottayasamy Seenivasagam (Other)
Responsible Party: Sponsor-Investigator, Rajkumar Kottayasamy Seenivasagam, MCh Surgical Oncology trainee, Government Royapettah Hospital
Organization: Government Royapettah Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRHCO-01
Record Dates: First submitted 2013-08-03; First posted 2013-08-07 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma Cervix
Keywords: Bulky cervical cancers; Neoadjuvant Chemotherapy; Neoadjuvant Chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Concurrent Radical Chemoradiation (Active Comparator): Paclitaxel(175 mg/sq.m) + Cisplatin (75 mg/sq.m) chemotherapy - 2 cycles of 3 weekly cycle Concurrent Radiotherapy - 50 Gy EBRT + Brachytherapy (7Gy HDR x 3 doses) All to be completed within 8-10 weeks
  Interventions: Drug: Chemotherapy; Radiation: External Beam Radiotherapy; Radiation: Brachytherapy
- Neoadjuvant Chemoradiation + Radical Hysterectomy (Experimental): Paclitaxel(175 mg/m2) + Cisplatin(75 mg/m2) chemotherapy - 2 cycles of 3 weekly cycle Concurrent Radiotherapy - 50 Gy EBRT - completed within 5 weeks Radical Hysterectomy - 3 weeks after completion of RT All to be completed within 8-10 weeks
  Interventions: Drug: Chemotherapy; Radiation: External Beam Radiotherapy; Procedure: Radical Hysterectomy
- Neoadjuvant Chemotherapy + Radical Hysterectomy (Experimental): Paclitaxel(175 mg/m2) + Cisplatin (75 mg/m2) chemotherapy - 3 cycles of 3 weekly cycle Radical Hysterectomy - 3 weeks after completion of chemotherapy All to be completed within 8-10 weeks
  Interventions: Drug: Chemotherapy; Procedure: Radical Hysterectomy

INTERVENTIONS:
Drug: Chemotherapy — cisplatin 75 mg/m2 Paclitaxel 175 mg/m2
Radiation: External Beam Radiotherapy — 50 Gy/2 Gy/25 # external beam RT to cervix. four field technique. given concurrently with chemotherapy weeks 1 - 5
  Arms: Concurrent Radical Chemoradiation; Neoadjuvant Chemoradiation + Radical Hysterectomy
Radiation: Brachytherapy — Ir - 192 HDR Brachytherapy - intracavitary. 7Gy x 3#. given after completion of chemoRT.
  Arms: Concurrent Radical Chemoradiation
Procedure: Radical Hysterectomy — Type III Radical Hysterectomy + Bilateral Pelvic Node Dissection
  Arms: Neoadjuvant Chemoradiation + Radical Hysterectomy; Neoadjuvant Chemotherapy + Radical Hysterectomy

SUMMARY:
The aim of this study is to establish the role of neoadjuvant chemotherapy and chemo irradiation in carcinoma cervix and to compare its results with the concurrent chemo irradiation in terms of overall survival, disease free survival and quality of life.

DETAILED DESCRIPTION:
Early stage bulky cancers of the cervix, (defined as FIGO Stages IB2, IIA2 and IIB) form a distinctive subset of "curable" cervical cancers with good 5 year survival rates with adequate treatment. Concurrent chemo radiation with or without salvage surgery is at present the standard of care for this group of cervical cancers. However, when pelvic recurrences occur, the morbidity of salvage surgery after radiotherapy, especially brachytherapy is often higher than the morbidity of salvage radiotherapy following radical surgery. The advantages of downsizing the disease without the use of brachytherapy are tempting and open a completely new philosophy in radical treatment for "curable" early stage bulky cancers of the cervix. This approach is appealing especially in developing countries where the load of cervical cancers is high and radiotherapy (brachytherapy) resources are scarce.

The results of two Phase II trials conducted at Govt. Royapettah Hospital, Chennai (Neoadjuvant Chemotherapy followed by Radical Hysterectomy: Cisplatin + 5FU vs. Cisplatin +Paclitaxel) and at Govt. General Hospital,Chennai (Neoadjuvant Chemoradiation with weekly cisplatin and 50 EBRT followed by radical Hysterectomy) and one retrospective study ( Preoperative 50 GY EBRT followed by Radical Hysterectomy) have shown similar response rates and acceptable toxicity profiles when compared to concurrent chemoradiation (EBRT + Brachytherapy+ Chemotherapy). Similar studies have been published elsewhere with similar results.

With this in mind we are planning to conduct a Phase III Randomised control trial comparing Neoadjuvant Chemotherapy + Radical Hysterectomy and Neoadjuvant Chemoradiation + Radical Hysterectomy with concurrent chemoradiation in this subset of cervical cancers

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed bulky cervical Squamous cell carcinoma (FIGO stage IB2, II A2, IIB).
2. Age 18-60 years
3. Karnofsky performance status of ≥70%; ECOG PS ≤ 2

Exclusion Criteria:

1. Nonsquamous Histologies
2. Other systemic diseases, comorbidities precluding full participation in the study
3. Concomitant treatment with any experimental drug
4. Pregnant or nursing women
5. Previous or concomitant malignant diseases other than non-melanoma skin cancer
6. Previous radiation to the pelvis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall and Disease free Survival | 3 year
Overall and Disease free Survival | 5 year

SECONDARY OUTCOMES:
Acute Adverse reactions and complications | Less than 10 weeks
SubAcute Adverse reactions and complications | 10 weeks - 6 months
Chronic Adverse reactions and complications | 6 months to 5 years

OTHER OUTCOMES:
Quality of Life | 3,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rajaraman Ramamurthy, MS MCh, Study Chair — centre for oncology, Government Royapettah Hospital
Locations (1):
- Government Royapettah Hospital, Chennai, Tamil Nadu, India